CLINICAL TRIAL: NCT04839341
Title: A Phase I, Open-labeled Multicenter Study to Determine Pharmacokinetics, Safety, Tolerability and Efficacy of Uproleselan in Combination With Chemotherapy in Chinese Patients With Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: Study to Evaluate PK and Safety With Uproleselan Combined With Chemotherapy to Treat Chinese R/R AML Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Apollomics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APL-106-01
Record Dates: First submitted 2021-03-22; First posted 2021-04-09 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Relapsed/Refractory AML
Keywords: AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — uproleselan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A Phase I, open-labeled multicenter study (Experimental): Uproleselan in combination with mitoxantrone, etoposide and cytarabine (MEC)
  Interventions: Drug: Uproleselan

INTERVENTIONS:
Drug: Uproleselan — A rationally designed E-selectin antagonist used to inhibit binding of cells to E-selectin
  Other Names: GMI-1271

SUMMARY:
This study will evaluate the safety and tolerability of uproleselan(GMI-1271), a specific E-selectin antagonist, and characterize the pharmacokinetic (PK) profile of uproleselan, in combination with chemotherapy to treat Chinese relapsed/refractory AML patients.

DETAILED DESCRIPTION:
This study is a multicenter open-labelled study conducted in subjects with relapsed or refractory AML in China. The study includes the following phases: screening phase, induction phase, consolidation phase baseline, consolidation phase and follow-up period.

Screening phase:

This study will enroll 12 subjects, who are 18 to 60 years (inclusive) at the time of signing the Informed Consent Form (ICF), and with the diagnosis as relapsed or refractory AML. Screening is conducted 21 days to 2 days before administration, and signed ICF by the subject must be obtained before screening.

Baseline period:

The baseline period is 1 day before study drug administration.

Induction treatment:

During the induction phase, subjects will receive 8 consecutive days of uproleselan treatment and 5 consecutive days of MEC (mitoxantrone, etoposide, and cytarabine combined regimen) chemotherapy.

Consolidation baseline:

The baseline of the consolidation phase is 1 day before the treatment administration of the consolidation phase.

Consolidation treatment:

Subjects who met the criteria for consolidation treatment started the consolidation period at the 29th day of the previous treatment cycle at the earliest and the 65th day at the latest.

Follow-up period:

Each subject should complete the following follow-up stage: (1) Response evaluation to determine remission to the induction treatment (induction period); (2) EOT assessment after completing the last consolidation treatment cycle; (3) Death. Survival and long-term follow-up, including initiation of new anti-leukemia treatment (within 6 months after the last uproleselan/placebo administration), recurrence, HSCT and survival events, monthly (±14 days) for 2 years after the end of treatment, and afterwards quarterly (±14 days). The longest survival follow-up time is 3 years (calculated from the start of treatment).

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years and ≤60 years in age
2. AML (including secondary AML) diagnosed as per WHO standards (2008).
3. For refractory AML, only cytarabine/daunorubicin(or Idarubicin) as can be applied repeatedly(maximal twice) as induction, no other chemotherapy are allowed to be applied Venatoclax /hypomethylation drug [HMA] can be used before and after chemotherapy.

   1. For relapse AML, it must be the first or second relapse, and remain untreated.
   2. Certain regimens (Venatoclax/HMA, Venetoclax/LDAC, HMA single agent) and FLT3 inhibitors, tyrosine kinase inhibitors, IDH1/IDH2 inhibitors or similar targeted inhibitors used alone are not considered cytotoxic chemotherapy are allowed.
4. ECOG performance status score is 0 to 2.
5. Stable hemodynamics and good organ function.

Exclusion Criteria:

1. Patients with acute promyelocytic leukemia, acute leukemia of ambiguous lineage (biphenotypic leukemia), chronic myeloid leukemia with myeloid blast crisis, or secondary refractory AML.
2. Active signs or symptoms of CNS involvement by malignancy.
3. Stem cell transplantation ≤4 months prior to dosing.
4. Any immunotherapy or radiotherapy therapy within 28 days of dosing; any other experimental therapy or chemotherapy within 14 days of dosing.
5. Prior use of G-CSF, CM-CSF or plerixafor within 7 days of dosing.
6. Inadequate organ function.
7. Abnormal liver function.
8. Known active infection with hepatitis A, B, or C, or human immunodeficiency virus.
9. Moderate kidney dysfunction (glomerular filtration rate <45 mL/min).
10. Uncontrolled acute life-threatening bacterial, viral, or fungal infection.
11. Clinically significant cardiovascular disease.
12. Major surgery within 4 weeks of dosing.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentration (Tmax) | 14 days
  To assess the pharmacokinetic profile in patients with relapsed/refractory AML.
Peak plasma concentration (Cmax) | 14 days
  To assess the pharmacokinetic profile in patients with relapsed/refractory AML.
Area under the plasma concentration-time curve from time zero to 12 hours (AUC0-12) | 14 days
  To assess the pharmacokinetic profile in patients with relapsed/refractory AML.
The area under the plasma concentration-time curve (AUC0-t) from time zero to the last measurable time point | 14 days
  To assess the pharmacokinetic profile in patients with relapsed/refractory AML.
The Incidence of Adverse Events | Up to 10 months
  Number of participants with an AE.
The tolerance of participants with relapsed/refractory AML. | Up to 10 months
  Number of participants could tolerate the Uproleselan combined with chemotherapy.

SECONDARY OUTCOMES:
OS | Up to 3 years
  Defined as the period from when the subject receives the first dose of the study drug to death from any cause;
Remission rate (rate of CR, CR/CRi and CR/CRh) | Up to 60 days
  Defined as the rate of subjects who reach CR, CR/CRi and CR/CRh;
CTCAE grade 3 and 4 oral mucositis | Up to 254 days
  The incidence of CTCAE grade 3 and 4 oral mucositis during the treatment duration.

CONTACTS AND LOCATIONS:
Overall Officials: Jianxiang Wang, PhD, Principal Investigator — Institute of Hematology and Blood Disease Hospital, Chinese Academy of Medical Sciences
Locations (2):
- China (2):
  - Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Zhejiang University, Hangzhou

IPD SHARING:
Plan to Share IPD: No